CLINICAL TRIAL: NCT04019093
Title: Acute Effects of Alcohol Use on Chronic Orofacial Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB201801911-N; R21AA026805 (NIH)
Record Dates: First submitted 2019-07-11; First posted 2019-07-15 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Temporomandibular Joint Disorders
Keywords: alcohol effects
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: People with and without jaw pain, including temporomandibular joint and muscle disorder (TMD) will receive an active oral dose of alcohol or placebo in a counterbalanced manner.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jaw pain patients (Experimental): Individuals seeking care for jaw pain, including temporomandibular joint and muscle disorder (TMD).
  Interventions: Drug: Ethanol; Other: Placebo
- Healthy controls (Experimental): Healthy social drinkers without jaw pain recruited as a comparison group.
  Interventions: Drug: Ethanol; Other: Placebo

INTERVENTIONS:
Drug: Ethanol — A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL.
Other: Placebo — A beverage that does not meaningfully increase breath alcohol concentration.

SUMMARY:
Self-medication of pain with alcohol is a common, yet risky, behavior among individuals with chronic orofacial pain. Chronic pain status may affect the degree to which alcohol use relieves pain, but the independent contributions of pain chronification and alcohol-related expectations and conditioning have not been previously studied. This project addresses this gap in knowledge and will inform further research and clinical/translational efforts for reducing risk associated with these behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Positive diagnosis of jaw pain, including temporomandibular joint and muscle disorder (TMD) (jaw pain group only)
* Consume at least 1 drink/month over the past 6 months

Exclusion Criteria:

* History of chronic pain other than jaw pain or TMD
* Current use of opioids
* Current major depression
* History of any psychotic disorder
* Undercontrolled hypertension or diabetes
* History of neurologic disease
* History of serious medical illness
* History of drug or alcohol dependence, including nicotine, or a pattern of hazardous alcohol use

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Boissoneault, PhD, Principal Investigator — University of Florida
Locations (1):
- Center for Pain Research and Behavioral Health at UF Health, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alexander C, Bush NJ, Neubert JK, Robinson M, Boissoneault J. Expectancy of alcohol analgesia moderates perception of pain relief following acute alcohol intake. Exp Clin Psychopharmacol. 2024 Apr;32(2):228-235. doi: 10.1037/pha0000664. Epub 2023 Jun 26. PMID 37358545

RESULTS

PARTICIPANT FLOW:
Groups:
- Jaw Pain Patients: Ethanol First, Then Placebo: Individuals seeking care for jaw pain, including temporomandibular joint and muscle disorder (TMD), randomized to receive ethanol first, followed by placebo.
  The first laboratory session lasted 4-8 hours, followed by a minimum 48 hour gap, and the second laboratory session lasted 4-8 hours.
  Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL.
  Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
- Healthy Controls: Ethanol First, Then Placebo: Healthy social drinkers without jaw pain recruited as a comparison group who received ethanol first, randomized to receive ethanol first, followed by placebo.
  The first laboratory session lasted 4-8 hours, followed by a minimum 48 hour gap, and the second laboratory session lasted 4-8 hours.
  Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL.
  Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
- Jaw Pain Patients: Placebo First, Then Ethanol: Individuals seeking care for jaw pain, including temporomandibular joint and muscle disorder (TMD), randomized to receive placebo first, followed by ethanol.
  The first laboratory session lasted 4-8 hours, followed by a minimum 48 hour gap, and the second laboratory session lasted 4-8 hours.
  Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL.
  Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
- Healthy Controls: Placebo First, Then Ethanol: Healthy social drinkers without jaw pain recruited as a comparison group who received ethanol first, randomized to receive placebo first, followed by ethanol.
  The first laboratory session lasted 4-8 hours, followed by a minimum 48 hour gap, and the second laboratory session lasted 4-8 hours.
  Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL.
  Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
Period: Overall Study
Arm/Group | Jaw Pain Patients: Ethanol First, Then Placebo | Healthy Controls: Ethanol First, Then Placebo | Jaw Pain Patients: Placebo First, Then Ethanol | Healthy Controls: Placebo First, Then Ethanol
Started | 9 | 16 | 10 | 13
Completed | 9 | 16 | 10 | 13
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Jaw Pain Patients | Healthy Controls | Total
Number analyzed (Participants) | 19 | 29 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.74 (5) | 25.72 (4.12) | 26.13 (4.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 36
  Male | 2 | 10 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 9 | 13
  Not Hispanic or Latino | 15 | 20 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 12 | 17 | 29
  More than one race | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 29 | 48
Alcohol Use Disorders Identification Test (total score) [Mean (Standard Deviation); unit: units on a scale] — The Alcohol Use Disorders Identification Test (AUDIT) is a standardized assessment of drinking frequency and heaviness, as well as consequences associated with alcohol intake. Higher scores reflect heavier/more frequent drinking and more severe alcohol-related consequences. Items are summed to compute total score, which can range from 0-40.
  units on a scale | 4.37 (1.77) | 4.31 (1.67) | 4.33 (1.69)
Quantity-Frequency Index [Mean (Standard Deviation); unit: oz. absolute ethanol consumed per day] | .426 (.35) | .551 (.39) | .48 (.36)
Max Quantity (oz. abs. EtOH) [Mean (Standard Deviation); unit: oz. absolute ethanol] | 4.29 (2.01) | 3.74 (1.41) | 3.96 (1.67)
Oral Health Impact Profile - TMDs (total score) [Mean (Standard Deviation); unit: units on a scale] — The Oral Health Impact Profile - TMDs is a temporomandibular joint and muscle disorder (TMD) specific version of the Oral Health Impact Profile. Total scores are generated by summing each item and range from 0-88. Higher scores indicate more severe TMD-related symptoms and quality of life impacts.
  units on a scale | 31.79 (14.74) | 10.14 (11.26) | 18.71 (16.53)

OUTCOME MEASURES:

1. Primary Outcome: Pressure Pain Threshold
Description: Pressure at which stimulation at the masseter insertion becomes painful, in lbf. Positive values represent higher pain thresholds.
Time Frame: Day 1; Day 2 (Laboratory sessions will be separated by at least 48 hours.)
Measure: Mean (Standard Deviation); unit: lbf
Groups:
- Jaw Pain Patients: Ethanol: Individuals seeking care for jaw pain, including temporomandibular joint and muscle disorder (TMD).
  Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL.
- Healthy Controls: Ethanol: Healthy social drinkers without jaw pain recruited as a comparison group.
  Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL.
  Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
- Jaw Pain Patients: Placebo: Individuals seeking care for jaw pain, including temporomandibular joint and muscle disorder (TMD).
  Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
- Healthy Controls: Placebo: Healthy social drinkers without jaw pain recruited as a comparison group.
  Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
Arm/Group | Jaw Pain Patients: Ethanol | Healthy Controls: Ethanol | Jaw Pain Patients: Placebo | Healthy Controls: Placebo
Number analyzed (Participants) | 19 | 29 | 19 | 29
lbf | 4.56 (1.08) | 5.27 (1.37) | 3.81 (0.84) | 4.51 (1.21)
Statistical Analysis 1: Comparison: Jaw Pain Patients: Ethanol vs Healthy Controls: Ethanol vs Jaw Pain Patients: Placebo vs Healthy Controls: Placebo; 2 (beverage condition: alcohol vs. placebo) X 2 (group: chronic pain vs. healthy control) mixed general linear model on pressure threshold. Here we report the results of the analysis of the beverage condition X group interaction; Test type: Superiority; p = .99, ANOVA; F(1,46) = .001
Statistical Analysis 2: Comparison: Jaw Pain Patients: Ethanol vs Healthy Controls: Ethanol vs Jaw Pain Patients: Placebo vs Healthy Controls: Placebo; 2 (beverage condition: alcohol vs. placebo) X 2 (group: chronic pain vs. healthy control) mixed general linear model on pressure threshold. Here we report the results of the analysis of the main effect of beverage condition; Test type: Superiority; p < .0001, ANOVA; F(1,46)=12.55
Statistical Analysis 3: Comparison: Jaw Pain Patients: Ethanol vs Healthy Controls: Ethanol vs Jaw Pain Patients: Placebo vs Healthy Controls: Placebo; 2 (beverage condition: alcohol vs. placebo) X 2 (group: chronic pain vs. healthy control) mixed general linear model on pressure threshold. Here we report the results of the analysis of the main effect of group; Test type: Superiority; p = .015, ANOVA; F(1,46)=6.32

2. Primary Outcome: Pressure Pain Intensity
Description: Pain ratings associated with 4, 5, or 6 pound-feet (lbf) of pressure applied to the insertion of the masseter. VAS (visual analogue scale) pain intensity ratings anchored from 0 ("no pain at all") to 100 ("most intense imaginable") were collected. Higher values represent higher pain intensity.
Time Frame: Day 1; Day 2 (Laboratory sessions will be separated by at least 48 hours.)
Population: Participant ratings from stimuli that were not within 0.5 lbf of the target pressure were excluded from analyses. This resulted in exclusion of 3 participants' data from this analysis.
Measure: Mean (Standard Deviation); unit: VAS units
Groups:
- Jaw Pain Patients: Ethanol, 4lbf: Individuals seeking care for jaw pain, including temporomandibular joint and muscle disorder (TMD).
  Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL.
  4lbf: Pressure applied to masseter insertion
- Healthy Controls: Ethanol, 4lbf: Healthy social drinkers without jaw pain recruited as a comparison group.
  Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL.
  Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
  4lbf: Pressure applied to masseter insertion
- Jaw Pain Patients: Placebo, 4lbf: Individuals seeking care for jaw pain, including temporomandibular joint and muscle disorder (TMD).
  Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
  4lbf: Pressure applied to masseter insertion
- Healthy Controls: Placebo, 4lbf: Healthy social drinkers without jaw pain recruited as a comparison group.
  Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
  4lbf: Pressure applied to masseter insertion
- Jaw Pain Patients: Ethanol, 5lbf: Individuals seeking care for jaw pain, including temporomandibular joint and muscle disorder (TMD).
  Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL.
  5lbf: Pressure applied to masseter insertion
- Healthy Controls: Ethanol, 5lbf: Healthy social drinkers without jaw pain recruited as a comparison group.
  Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL.
  Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
  5lbf: Pressure applied to masseter insertion
- Jaw Pain Patients: Placebo, 5lbf: Individuals seeking care for jaw pain, including temporomandibular joint and muscle disorder (TMD).
  Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
  5lbf: Pressure applied to masseter insertion
- Healthy Controls: Placebo, 5lbf: Healthy social drinkers without jaw pain recruited as a comparison group.
  Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
  5lbf: Pressure applied to masseter insertion
- Jaw Pain Patients: Ethanol, 6lbf: Individuals seeking care for jaw pain, including temporomandibular joint and muscle disorder (TMD).
  Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL.
  6lbf: Pressure applied to masseter insertion
- Healthy Controls: Ethanol, 6lbf: Healthy social drinkers without jaw pain recruited as a comparison group.
  Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL.
  Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
  6lbf: Pressure applied to masseter insertion
- Jaw Pain Patients: Placebo, 6lbf: Individuals seeking care for jaw pain, including temporomandibular joint and muscle disorder (TMD).
  Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
  6lbf: Pressure applied to masseter insertion
- Healthy Controls: Placebo, 6lbf: Healthy social drinkers without jaw pain recruited as a comparison group.
  Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
  6lbf: Pressure applied to masseter insertion
Arm/Group | Jaw Pain Patients: Ethanol, 4lbf | Healthy Controls: Ethanol, 4lbf | Jaw Pain Patients: Placebo, 4lbf | Healthy Controls: Placebo, 4lbf | Jaw Pain Patients: Ethanol, 5lbf | Healthy Controls: Ethanol, 5lbf | Jaw Pain Patients: Placebo, 5lbf | Healthy Controls: Placebo, 5lbf | Jaw Pain Patients: Ethanol, 6lbf | Healthy Controls: Ethanol, 6lbf | Jaw Pain Patients: Placebo, 6lbf | Healthy Controls: Placebo, 6lbf
Number analyzed (Participants) | 17 | 28 | 17 | 28 | 17 | 28 | 17 | 28 | 17 | 28 | 17 | 28
VAS units | 23.96 (28.03) | 12.76 (13.44) | 32.39 (19.95) | 22.05 (17.72) | 35.43 (19.67) | 20.92 (17.02) | 41.81 (20.28) | 29.98 (23.89) | 37.19 (23.90) | 26.95 (23.06) | 46.10 (22.97) | 34.03 (22.94)
Statistical Analysis 1: Comparison: Jaw Pain Patients: Ethanol, 4lbf vs Healthy Controls: Ethanol, 4lbf vs Jaw Pain Patients: Placebo, 4lbf vs Healthy Controls: Placebo, 4lbf vs Jaw Pain Patients: Ethanol, 5lbf vs Healthy Controls: Ethanol, 5lbf vs Jaw Pain Patients: Placebo, 5lbf vs Healthy Controls: Placebo, 5lbf vs Jaw Pain Patients: Ethanol, 6lbf vs Healthy Controls: Ethanol, 6lbf vs Jaw Pain Patients: Placebo, 6lbf vs Healthy Controls: Placebo, 6lbf; 2 (beverage condition: alcohol vs. placebo) X 2 (group: chronic pain vs. healthy control) x 2 (pressure level: 4 lbf vs. 5 lbf vs 6 lbf) mixed general linear model on pain intensity. Here we report the results of the analysis of the pressure level X group interaction; Test type: Superiority; p = .76, ANOVA; F(2,82)=.20
Statistical Analysis 2: Comparison: Jaw Pain Patients: Ethanol, 4lbf vs Healthy Controls: Ethanol, 4lbf vs Jaw Pain Patients: Placebo, 4lbf vs Healthy Controls: Placebo, 4lbf vs Jaw Pain Patients: Ethanol, 5lbf vs Healthy Controls: Ethanol, 5lbf vs Jaw Pain Patients: Placebo, 5lbf vs Healthy Controls: Placebo, 5lbf vs Jaw Pain Patients: Ethanol, 6lbf vs Healthy Controls: Ethanol, 6lbf vs Jaw Pain Patients: Placebo, 6lbf vs Healthy Controls: Placebo, 6lbf; 2 (beverage condition: alcohol vs. placebo) X 2 (group: chronic pain vs. healthy control) x 2 (pressure level: 4 lbf vs. 5 lbf vs 6 lbf) mixed general linear model on pain intensity. Here we report the results of the analysis of the pressure level X beverage condition interaction; Test type: Superiority; p = .52, ANCOVA; F(2,82)=.66
Statistical Analysis 3: Comparison: Jaw Pain Patients: Ethanol, 4lbf vs Healthy Controls: Ethanol, 4lbf vs Jaw Pain Patients: Placebo, 4lbf vs Healthy Controls: Placebo, 4lbf vs Jaw Pain Patients: Ethanol, 5lbf vs Healthy Controls: Ethanol, 5lbf vs Jaw Pain Patients: Placebo, 5lbf vs Healthy Controls: Placebo, 5lbf vs Jaw Pain Patients: Ethanol, 6lbf vs Healthy Controls: Ethanol, 6lbf vs Jaw Pain Patients: Placebo, 6lbf vs Healthy Controls: Placebo, 6lbf; 2 (beverage condition: alcohol vs. placebo) X 2 (group: chronic pain vs. healthy control) x 2 (pressure level: 4 lbf vs. 5 lbf vs 6 lbf) mixed general linear model on pain intensity. Here we report the results of the analysis of the main effect of beverage condition; Test type: Superiority; p = .04, ANOVA; F(1,41)=4.53, p=.04
Statistical Analysis 4: Comparison: Jaw Pain Patients: Ethanol, 4lbf vs Healthy Controls: Ethanol, 4lbf vs Jaw Pain Patients: Placebo, 4lbf vs Healthy Controls: Placebo, 4lbf vs Jaw Pain Patients: Ethanol, 5lbf vs Healthy Controls: Ethanol, 5lbf vs Jaw Pain Patients: Placebo, 5lbf vs Healthy Controls: Placebo, 5lbf vs Jaw Pain Patients: Ethanol, 6lbf vs Healthy Controls: Ethanol, 6lbf vs Jaw Pain Patients: Placebo, 6lbf vs Healthy Controls: Placebo, 6lbf; 2 (beverage condition: alcohol vs. placebo) X 2 (group: chronic pain vs. healthy control) x 2 (pressure level: 4 lbf vs. 5 lbf vs 6 lbf) mixed general linear model on pain intensity. Here we report the results of the analysis of the main effect of group; Test type: Superiority; p = .017, ANOVA; F(1,41)=6.24
Statistical Analysis 5: Comparison: Jaw Pain Patients: Ethanol, 4lbf vs Healthy Controls: Ethanol, 4lbf vs Jaw Pain Patients: Placebo, 4lbf vs Healthy Controls: Placebo, 4lbf vs Jaw Pain Patients: Ethanol, 5lbf vs Healthy Controls: Ethanol, 5lbf vs Jaw Pain Patients: Placebo, 5lbf vs Healthy Controls: Placebo, 5lbf vs Jaw Pain Patients: Ethanol, 6lbf vs Healthy Controls: Ethanol, 6lbf vs Jaw Pain Patients: Placebo, 6lbf vs Healthy Controls: Placebo, 6lbf; 2 (beverage condition: alcohol vs. placebo) X 2 (group: chronic pain vs. healthy control) x 2 (pressure level: 4 lbf vs. 5 lbf vs 6 lbf) mixed general linear model on pain intensity. Here we report the results of the analysis of the main effect of pressure level; Test type: Superiority; p < .0001, ANOVA; F(2,82)=48.41

3. Primary Outcome: Perceived Relief
Description: Ratings of relief from pain associated with consumption of the study beverage following application of 4, 5, or 6 lbf stimuli. VAS (visual analogue scale) assessing perceived relief anchored from 0 ("No relief at all") to 100 ("Most profound relief imaginable"). Higher values represent greater perceived relief.
Time Frame: Day 1; Day 2 (Laboratory sessions will be separated by at least 48 hours.)
Population: One participant had missing data on this measure, resulting from exclusion from analyses.
Measure: Mean (Standard Deviation); unit: VAS units
Arm/Group | Jaw Pain Patients: Ethanol, 4lbf | Healthy Controls: Ethanol, 4lbf | Jaw Pain Patients: Placebo, 4lbf | Healthy Controls: Placebo, 4lbf | Jaw Pain Patients: Ethanol, 5lbf | Healthy Controls: Ethanol, 5lbf | Jaw Pain Patients: Placebo, 5lbf | Healthy Controls: Placebo, 5lbf | Jaw Pain Patients: Ethanol, 6lbf | Healthy Controls: Ethanol, 6lbf | Jaw Pain Patients: Placebo, 6lbf | Healthy Controls: Placebo, 6lbf
Number analyzed (Participants) | 19 | 28 | 19 | 28 | 19 | 28 | 19 | 28 | 19 | 28 | 19 | 28
VAS units | 40.58 (31.31) | 39.79 (30.58) | 7.91 (13.71) | 5.51 (11.36) | 41.00 (28.27) | 42.75 (30.14) | 7.20 (13.01) | 5.57 (11.13) | 39.72 (30.05) | 43.65 (29.61) | 7.20 (13.41) | 5.89 (13.11)
Statistical Analysis 1: Comparison: Jaw Pain Patients: Ethanol, 4lbf vs Healthy Controls: Ethanol, 4lbf vs Jaw Pain Patients: Placebo, 4lbf vs Healthy Controls: Placebo, 4lbf vs Jaw Pain Patients: Ethanol, 5lbf vs Healthy Controls: Ethanol, 5lbf vs Jaw Pain Patients: Placebo, 5lbf vs Healthy Controls: Placebo, 5lbf vs Jaw Pain Patients: Ethanol, 6lbf vs Healthy Controls: Ethanol, 6lbf vs Jaw Pain Patients: Placebo, 6lbf vs Healthy Controls: Placebo, 6lbf; 2 (beverage condition: alcohol vs. placebo) X 2 (group: chronic pain vs. healthy control) x 2 (pressure level: 4 lbf vs. 5 lbf vs 6 lbf) mixed general linear model on pain relief. Here we report the results of the analysis of the beverage condition X pressure level X group interaction; Test type: Superiority; p = .50, ANOVA; F (2, 82) = 0.69
Statistical Analysis 2: Comparison: Jaw Pain Patients: Ethanol, 4lbf vs Healthy Controls: Ethanol, 4lbf vs Jaw Pain Patients: Placebo, 4lbf vs Healthy Controls: Placebo, 4lbf vs Jaw Pain Patients: Ethanol, 5lbf vs Healthy Controls: Ethanol, 5lbf vs Jaw Pain Patients: Placebo, 5lbf vs Healthy Controls: Placebo, 5lbf vs Jaw Pain Patients: Ethanol, 6lbf vs Healthy Controls: Ethanol, 6lbf vs Jaw Pain Patients: Placebo, 6lbf vs Healthy Controls: Placebo, 6lbf; 2 (beverage condition: alcohol vs. placebo) X 2 (group: chronic pain vs. healthy control) x 2 (pressure level: 4 lbf vs. 5 lbf vs 6 lbf) mixed general linear model on pain relief. Here we report the results of the analysis of the beverage condition X pressure level interaction; Test type: Superiority; p = .21, ANOVA; F(2,82)=1.58
Statistical Analysis 3: Comparison: Jaw Pain Patients: Ethanol, 4lbf vs Healthy Controls: Ethanol, 4lbf vs Jaw Pain Patients: Placebo, 4lbf vs Healthy Controls: Placebo, 4lbf vs Jaw Pain Patients: Ethanol, 5lbf vs Healthy Controls: Ethanol, 5lbf vs Jaw Pain Patients: Placebo, 5lbf vs Healthy Controls: Placebo, 5lbf vs Jaw Pain Patients: Ethanol, 6lbf vs Healthy Controls: Ethanol, 6lbf vs Jaw Pain Patients: Placebo, 6lbf vs Healthy Controls: Placebo, 6lbf; 2 (beverage condition: alcohol vs. placebo) X 2 (group: chronic pain vs. healthy control) x 2 (pressure level: 4 lbf vs. 5 lbf vs 6 lbf) mixed general linear model on pain relief. Here we report the results of the analysis of the pressure level X group interaction; Test type: Superiority; p = .053, ANOVA; F(2,82)=3.06
Statistical Analysis 4: Comparison: Jaw Pain Patients: Ethanol, 4lbf vs Healthy Controls: Ethanol, 4lbf vs Jaw Pain Patients: Placebo, 4lbf vs Healthy Controls: Placebo, 4lbf vs Jaw Pain Patients: Ethanol, 5lbf vs Healthy Controls: Ethanol, 5lbf vs Jaw Pain Patients: Placebo, 5lbf vs Healthy Controls: Placebo, 5lbf vs Jaw Pain Patients: Ethanol, 6lbf vs Healthy Controls: Ethanol, 6lbf vs Jaw Pain Patients: Placebo, 6lbf vs Healthy Controls: Placebo, 6lbf; 2 (beverage condition: alcohol vs. placebo) X 2 (group: chronic pain vs. healthy control) x 2 (pressure level: 4 lbf vs. 5 lbf vs 6 lbf) mixed general linear model on pain relief. Here we report the results of the analysis of the beverage condition X group interaction; Test type: Superiority; p = .98, ANOVA; F(1,41)=.001
Statistical Analysis 5: Comparison: Jaw Pain Patients: Ethanol, 4lbf vs Healthy Controls: Ethanol, 4lbf vs Jaw Pain Patients: Placebo, 4lbf vs Healthy Controls: Placebo, 4lbf vs Jaw Pain Patients: Ethanol, 5lbf vs Healthy Controls: Ethanol, 5lbf vs Jaw Pain Patients: Placebo, 5lbf vs Healthy Controls: Placebo, 5lbf vs Jaw Pain Patients: Ethanol, 6lbf vs Healthy Controls: Ethanol, 6lbf vs Jaw Pain Patients: Placebo, 6lbf vs Healthy Controls: Placebo, 6lbf; 2 (beverage condition: alcohol vs. placebo) X 2 (group: chronic pain vs. healthy control) x 2 (pressure level: 4 lbf vs. 5 lbf vs 6 lbf) mixed general linear model on pain relief. Here we report the results of the analysis of the main effect of pressure level; Test type: Superiority; p = .71, ANOVA; F(2,82)=.34
Statistical Analysis 6: Comparison: Jaw Pain Patients: Ethanol, 4lbf vs Healthy Controls: Ethanol, 4lbf vs Jaw Pain Patients: Placebo, 4lbf vs Healthy Controls: Placebo, 4lbf vs Jaw Pain Patients: Ethanol, 5lbf vs Healthy Controls: Ethanol, 5lbf vs Jaw Pain Patients: Placebo, 5lbf vs Healthy Controls: Placebo, 5lbf vs Jaw Pain Patients: Ethanol, 6lbf vs Healthy Controls: Ethanol, 6lbf vs Jaw Pain Patients: Placebo, 6lbf vs Healthy Controls: Placebo, 6lbf; 2 (beverage condition: alcohol vs. placebo) X 2 (group: chronic pain vs. healthy control) x 2 (pressure level: 4 lbf vs. 5 lbf vs 6 lbf) mixed general linear model on pain relief. Here we report the results of the analysis of the main effect of group; Test type: Superiority; p = .71, ANOVA; F(1,41)=.14
Statistical Analysis 7: Comparison: Jaw Pain Patients: Ethanol, 4lbf vs Healthy Controls: Ethanol, 4lbf vs Jaw Pain Patients: Placebo, 4lbf vs Healthy Controls: Placebo, 4lbf vs Jaw Pain Patients: Ethanol, 5lbf vs Healthy Controls: Ethanol, 5lbf vs Jaw Pain Patients: Placebo, 5lbf vs Healthy Controls: Placebo, 5lbf vs Jaw Pain Patients: Ethanol, 6lbf vs Healthy Controls: Ethanol, 6lbf vs Jaw Pain Patients: Placebo, 6lbf vs Healthy Controls: Placebo, 6lbf; 2 (beverage condition: alcohol vs. placebo) X 2 (group: chronic pain vs. healthy control) x 2 (pressure level: 4 lbf vs. 5 lbf vs 6 lbf) mixed general linear model on pain relief. Here we report the results of the analysis of the main effect of beverage condition; Test type: Superiority; p < .0001, ANOVA; F(1,41)=55.02

ADVERSE EVENTS:
Time Frame: Duration of study participation (4-8 hours per study session, with at least 48 hours separating each session)
Groups:
- Jaw Pain Patients: Ethanol; Jaw Pain Patients: Placebo: Individuals seeking care for jaw pain, including temporomandibular joint and muscle disorder (TMD).
  Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL.
  Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
- Healthy Controls: Placebo: Healthy social drinkers without jaw pain recruited as a comparison group.
  Ethanol: A beverage containing dose of ethanol individually determined to raise a participant's breath alcohol concentration up to approximately 0.08 g/dL.
  Placebo: A beverage that does not meaningfully increase breath alcohol concentration.
Arm/Group | Jaw Pain Patients: Ethanol | Healthy Controls: Ethanol | Jaw Pain Patients: Placebo | Healthy Controls: Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/29 | 0/19 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/29 | 0/19 | 0/29
Other Adverse Events (participants affected / at risk) | 0/19 | 1/29 | 0/19 | 0/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Jaw Pain Patients: Ethanol (N=19) | Healthy Controls: Ethanol (N=29) | Jaw Pain Patients: Placebo (N=19) | Healthy Controls: Placebo (N=29)
Nausea and vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Approximately 2.5 hours after consuming the study beverage, while metabolizing alcohol dose prior to transport home, participant reported feeling nauseous and vomited. Participant's BrAC was 0.04.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT04019093/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/93/NCT04019093/ICF_001.pdf